CLINICAL TRIAL: NCT01763710
Title: Neurotoxicity Characterization Phase II Randomized Study of Nab-paclitaxel Versus Conventional Paclitaxel as First-line Therapy of Metastatic HER2-negative Breast Cancer.
Brief Title: Neurotoxicity Characterization Study of Nab-paclitaxel Versus Conventional Paclitaxel in Metastatic Breast Cancer
Acronym: neurabrax
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Oncosur (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ONCOSUR-2012-01
Record Dates: First submitted 2012-12-14; First posted 2013-01-09 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Neurotoxicity
MeSH Terms: conditions — Breast Neoplasms; Neurotoxicity Syndromes | interventions — Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Active Comparator): Paclitaxel 80 mg/m2 days 1, 8 and 15
  Interventions: Drug: Paclitaxel 80 mg/m2
- Arm B (Experimental): Nab-paclitaxel 100 mg/m2 days 1, 8 and 15
  Interventions: Drug: Nab-paclitaxel 100 mg/m2 days 1, 8 and 15
- Arm C (Experimental): Nab-paclitaxel 150 mg/m2 days 1, 8 and 15
  Interventions: Drug: Nab-paclitaxel 150 mg/m2 days 1, 8 and 15
- Arm D (Experimental): Nab-paclitaxel 150 mg/m2 days 1 and 15
  Interventions: Drug: Nab-paclitaxel 150 mg/m2 days 1 and 15

INTERVENTIONS:
Drug: Paclitaxel 80 mg/m2 — Paclitaxel 80 mg/m2 days 1, 8 and 15
  Arms: Arm A
Drug: Nab-paclitaxel 100 mg/m2 days 1, 8 and 15 — Nab-paclitaxel 100 mg/m2 days 1, 8 and 15
  Arms: Arm B
Drug: Nab-paclitaxel 150 mg/m2 days 1, 8 and 15 — Nab-paclitaxel 150 mg/m2 days 1, 8 and 15
  Arms: Arm C
Drug: Nab-paclitaxel 150 mg/m2 days 1 and 15 — Nab-paclitaxel 150 mg/m2 days 1 and 15
  Arms: Arm D

SUMMARY:
Nanomedicines are currently being developed in the treatment of cancer due to their pharmacological advantages over traditional formulations; they provide a shorter infusion time and lower risks of hypersensitivity reactions associated with commonly used solvents.

Nab-paclitaxel is a nanoparticle albumin-bound particle form of paclitaxel that is thought to exploit natural albumin pathways to enhance the selective uptake and accumulation of paclitaxel at the site of the tumour, thus reducing its diffusion to normal tissues.

Nab-paclitaxel has been approved for the treatment of metastatic breast cancer patients who have failed first-line treatment for metastatic disease and for whom standard, anthracycline-containing therapy is not indicated.

SPARC is a cysteine rich acid protein that is overexpressed in a broad proportion of solid tumours. Expression of this protein could sensitize tumour cells to antitumor activity of Nab-paclitaxel, due to its union through albumin-binding to this protein.

First-line clinical trials have been developed with different Nab-paclitaxel regimens and also in combination with different chemotherapies and trastuzumab, showing a high level of efficacy.

Toxicity profile of Nab-paclitaxel is well characterized with significantly less haematological toxicities compared with conventional paclitaxel.

Nab-paclitaxel derived grade III neuropathy is short-lasting and more reversible than conventional paclitaxel-derived neuropathy, probably due to absence of Cremophor solvent, or due to paclitaxel itself.

However there is still a lack of clinical and physiological characterisation of Nab-paclitaxel induced neuropathy.

The current used tools for early detection and continuous evaluation of neurotoxicity are not optimal. Most used toxicity scales are limited, as they do not provide a detailed information of the severity of the neuropathy, its impact on quality of life, or physiopathology mechanisms.

In addition, an inter-individual variability exists in terms of neurotoxicity predisposition when taxanes are used; it could be related to polymorphic differences in genes implicated in transport and metabolism of these drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Women with histologically or cytologically of stage IV breast cancer.
2. Non-candidate patient to trastuzumab or lapatinib treatment as not presenting HER2 oncogene amplification.
3. Metastatic disease not previously treated with chemotherapy. It is allowed pre-treatment hormone with anti-target or bisphosphonates for advanced disease.
4. Measurable or evaluable disease by RECIST criteria.
5. Previous sensory neuropathy <= grade 1, according to NCI-CTCAE criteria, due to any reason.
6. Age> 18 years.
7. Performance status <2 (ECOG).
8. At least 12 months after the completion of adjuvant chemotherapy with taxanes to diagnosis of metastatic disease.
9. Creatinine <= 1.5mg/dL, AST (SGOT), ALT (SGPT) and alkaline phosphatase <= 2.5 x ULN (hepatic metastases absent) in the 14 days prior to study entry.
10. Hemoglobin> 10g/dl, WBC> 3000/mm3, platelets> 100000/mm3 and bilirubin <1.5 mg / dL in the 14 days prior to study entry.
11. Women of childbearing potential with negative pregnancy test within 14 days prior to study treatment.
12. Patients using adequate contraception throughout the entire duration of the study and until 4 weeks after completion of treatment.
13. At least 4 weeks after radiotherapy or major surgery, with complete recovery.
14. Life expectancy greater than 12 weeks.
15. Patients who are able to meet the requirements of the protocol.
16. Patients able to provide with two plasma samples (each sample 5cc) for analyzing polymorphisms.
17. Written informed consent.

Exclusion Criteria:

1. Prior chemotherapy treatment for metastatic disease.
2. Brain metastases.
3. Concomitant treatment with hormone therapy or immunotherapy for breast cancer, or during the two weeks prior to inclusion in the study.
4. Any concomitant medical or psychiatric illness including active infection.
5. History of any malignancy other than breast cancer in the past 5 years except carcinoma or basal cell skin carcinoma or carcinoma in situ of cervix.
6. Prior treatment with an investigational drug within the last 2 weeks.
7. Known hypersensitivity to paclitaxel or Cremophor.
8. Pregnant or breastfeeding.
9. Have any acute, subacute or chronic peripheral nerve or spinal cord in grade, at the time of inclusion, greater than or equal to 2 (NCI CTCAE v4.0).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
TNS - Total Neuropathy Score | Every 3 months up to 6 months

SECONDARY OUTCOMES:
Evaluate the incidence of neuropathy induced by study treatment (conventional paclitaxel vs nab-paclitaxel) | Every 3 weeks up to 24 weeks
Evaluate the electromyographic abnormalities and the correlation of these alterations with the assessment of the TNS scale and NCI-CTCAE (Common Toxicity Criteria for Adverse Effects) v4.0 | Every 12 weeks up to 24 weeks
Determine the predictive value of genetic variants (SNPs) for the development of neuropathy | In the two weeks before start treatment
Determine the clinical activity of both treatments (response rate, time to progression) | Every 8-12 weeks up to 24 weeks
Determine toxicity profile and safety of study treatments (NCI-CTCAE v4.0) | Every 2 weeks up to 24 weeks
Determine time to neurotoxicity onset | Every 2 weeks up to 24 weeks
Determine time to recovery from neurotoxicity | Every 2 weeks up to 24 weeks
Determine time to progression | Every 8-12 weeks up to 24 weeks
Assess quality of live (EORTC QLQ-C30 and EORTC QLQ-CIPN20) | Every 4 weeks up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ciruelos, MD, Study Director — Hospital 12 de Octubre, Servicio de Oncología Médica; Noelia Martínez, MD, Principal Investigator — Hoapital Ramón y Cajal, Servicio de Oncología Médica; Rafael Carrión, MD, Principal Investigator — Hospital Universitario del Sureste, Servicio de Oncología Médica; José A García Sáenz, MD, Principal Investigator — Hospital Clínico San Carlos, Servicio de Oncología Médica; María Echarri, Md, Principal Investigator — Hospital Universitario Severo Ochoa, Servicio de Oncología Médica; Blanca Cantos, MD, Principal Investigator — Hospital Universitario Puerta de hierro Majadahonda, Servicio de Oncología Médica; Coralía Bueno, MD, Principal Investigator — Hospital Universitario Infanta Cristina, Servicio de Oncología Médica; Miguel A Lara, MD, Principal Investigator — Hospital Universitario Infanta Leonor; Santos Enrech, MD, Principal Investigator — Hospital Universitario de Getafe, Servicio de Oncología Médica; Juan A Guerra, MD, Principal Investigator — Hospital Universitario de Fuenlabrada
Locations (10):
- Spain (10):
  - Hospital Universitario Del Sureste, Arganda, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Infanta Leonor, Madrid, Madrid
  - Hospital Ramón Y Cajal, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Infanta Cristina, Parla, Madrid

REFERENCES:
- [Derived] Ciruelos E, Apellaniz-Ruiz M, Cantos B, Martinez-Janez N, Bueno-Muino C, Echarri MJ, Enrech S, Guerra JA, Manso L, Pascual T, Dominguez C, Gonzalo JF, Sanz JL, Rodriguez-Antona C, Sepulveda JM. A Pilot, Phase II, Randomized, Open-Label Clinical Trial Comparing the Neurotoxicity of Three Dose Regimens of Nab-Paclitaxel to That of Solvent-Based Paclitaxel as the First-Line Treatment for Patients with Human Epidermal Growth Factor Receptor Type 2-Negative Metastatic Breast Cancer. Oncologist. 2019 Nov;24(11):e1024-e1033. doi: 10.1634/theoncologist.2017-0664. Epub 2019 Apr 25. PMID 31023863